CLINICAL TRIAL: NCT05732181
Title: The Role of 5% Lidocaine Patches in the Pain Control of Hepatocellular Carcinoma Patients Receiving Radiofrequency Ablation: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: The Role of 5% Lidocaine Patches in the Pain Control of Hepatocellular Carcinoma Patients Receiving Radiofrequency Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-ER-106-060
Record Dates: First submitted 2023-01-05; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-12

CONDITIONS: Liver Cancer; Post Ablation Syndrome
Keywords: Hepatocellular carcinoma; Radiofrequency ablation; Lidocaine patch
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine patch (Experimental)
  Interventions: Drug: The skin lidocaine patch.; Drug: Placebo
- Placebo (No Intervention)

INTERVENTIONS:
Drug: The skin lidocaine patch. — The skin patch is applied before RFA while admission and is changed every day till discharge. Pain severity is evaluated by visual analogue scale using a 10-point scale recorded before RFA and after the procedure.
  Arms: Lidocaine patch
Drug: Placebo — patch without drugs
  Arms: Lidocaine patch

SUMMARY:
Background: This study aims to test whether 5% lidocaine patches can reduce Radiofrequency ablation-induced pain. Methods: The study will enroll patients with hepatocellular carcinoma and schedule a radiofrequency ablation procedure. 200 patients will be invited to allocate randomly into study or control groups: pretreatment with a 5% lidocaine patch (LidotopⓇ) (Group A); pretreatment with a placebo patch (Group B); The skin patch is applied before Radiofrequency ablation (RFA) while admission, and is changed every day till discharge. Pain severity is evaluated by a visual analog scale using a 10-point scale recorded by a study nurse before RFA and after the procedure. The demographic data, hepatocellular carcinoma characteristics, analgesics usage, patient satisfaction with pain control, and visual analog scale will be compared between the two groups. Anticipated results: Pretreatment with 5% lidocaine patches is an effective and straight method of reducing Radiofrequency ablation-induced pain to reduce analgesics usage and improve patient satisfaction with pain control.

ELIGIBILITY:
Inclusion Criteria:

1. Adults diagnosed with liver cancer (HCC) by a physician and eligible for radiofrequency cautery (RFA).
2. Age is > = 18 years.
3. Whether there is cirrhosis combined with cirrhosis, the child-pugh score of those with cirrhosis must score < 8 points.
4. Communicative and able to express pain sensations.

Exclusion Criteria:

1. Those who are allergic to Lidocaine.
2. Those who suffer from skin diseases or have wounds on the abdomen that cannot be patched.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Pain severity | two days to three days.
  visual analogue scale using a 10-point scale recorded

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan